CLINICAL TRIAL: NCT05070221
Title: Safety and Efficacy Study of Oncolytic Virus（Intratumoral Injection）in Combination With HX-008（Intravenous Injection）and Axitinib in Melanoma Patients With Liver Metastasis Who Lack or Become Refractory to Standard Treatment
Brief Title: Study of Oncolytic Virus in Combination With HX-008 and Axitinib in Melanoma Patients With Liver Metastasis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Vice President, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH-OH2-014
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Melanoma Stage IV
MeSH Terms: conditions — Melanoma | interventions — Injections; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Patients histologically confirmed mucosal melanoma will get OH2 （once every two weeks）and HX-008 (once every three weeks)and Axitinib (once every day).
  Interventions: Drug: Recombinant Oncolytic HSV-2 Therapeutic Injecta (Vero Cell) for Human Use (rHSV2hGM-CSF); Drug: Recombinant humanized anti-PD-1 monoclonal antibody for injection; Drug: Axitinib
- Arm B (Experimental): Patients histologically confirmed non-mucosal melanoma will get OH2 （once every two weeks）and HX-008 (once every three weeks)and Axitinib (once every day).
  Interventions: Drug: Recombinant Oncolytic HSV-2 Therapeutic Injecta (Vero Cell) for Human Use (rHSV2hGM-CSF); Drug: Recombinant humanized anti-PD-1 monoclonal antibody for injection; Drug: Axitinib

INTERVENTIONS:
Drug: Recombinant Oncolytic HSV-2 Therapeutic Injecta (Vero Cell) for Human Use (rHSV2hGM-CSF) — less than 8mL/time，Q2W，i.t.；
  Other Names: OH2
Drug: Recombinant humanized anti-PD-1 monoclonal antibody for injection — 200mg/time，Q3W，i.v.；
  Other Names: HX-008
Drug: Axitinib — 5mg，bid，p.o.；
  Other Names: Inlyta®

SUMMARY:
Malignant melanoma, is a kind of malignant tumor derived from melanocytes. It is common in skin, mucous membrane, eye choroid and other parts. Melanoma is one of the fastest growing malignant tumors with an annual incidence rate of 3-5%. In 2012, there were 232000 new cases of melanoma and 55000 deaths worldwide. Though, the incidence rate of melanoma is relatively low in China, it has been increasing rapidly in recent years. Melanoma has seriously endangering the health of Chinese people.

Patients with stage Ⅳ melanoma have a poor prognosis. According to statistics, the median survival time of stage M1a melanoma is 15 months, while stage M1b is 8 months. The median survival time of bone metastasis melanoma is 6 months, while liver and brain metastasis is 4 months. The overall median survival time of metastatic melanoma is only 7.5 months, and the 2-year survival rate is 15%.

For patients with advanced melanoma, dacarbazine is the only chemotherapy drug approved by NMPA, but its overall effective rate is only 13.4%, and the median survival time is 5.6 ~ 11 months.

Therapies(new drugs or new combination treatments)with higher remission rate and longer survival are urgently needed for patients with advanced melanoma.

DETAILED DESCRIPTION:
This study is a single-center, non-randomized,open-label study to evaluate safety and efficacy of recombinant human GM-CSF herpes simplex virus（intratumoral injection） in combination with recombinant humanized anti-PD-1 monoclonal antibody (intravenous injection) and Axitinib for liver metastasis in stage IV melanoma.

This study is planned to enroll 30-45 patients with stage IV liver metastasis melanoma who lack or become refractory to standard treatment.

This study set scientific inclusion/exclusion criteria. Patients could be included in the group for treatment only after being strictly reviewed by researcher. The clinical research associate(CRA) will regularly monitor the research data during the whole study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign Informed Consent Form（ICF）, understand the study, be willing to follow and be able to complete all test procedures;
2. Male and female, 18-75 years old (including boundary value);
3. Histologically confirmed stage IV melanoma with liver metastasis who lacks or becomes refractory to standard treatment;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status is 0 or 1;
5. Expected survival at least 3 months;
6. The interval between the first administration and previous treatment (including chemotherapy, radiotherapy, targeted therapy, immunotherapy and biotherapy for melanoma) in the past is over 4 weeks, and has recovered to grade 1 from the adverse reactions of previous treatment;
7. At least one measurable or evaluable lesion;
8. Liver metastasis has lesions suitable for intratumoral injection;
9. Asymptomatic central nervous system metastasis or asymptomatic brain metastasis after treatment must be confirmed by CT / MRI that there is no disease progression, stable for at least 3 months, and no steroid treatment for at least 4 weeks;
10. Appropriate organs and hematopoietic function according to the following laboratory tests: neutrophil absolute count (neut#) ≥ 2.0 × 109/L； Absolute white blood cell count (WBC) ≥ 3.0 × 109/L； Platelet ≥ 100 × 109/L； Hemoglobin ≥ 90g / L; Serum creatinine ≤ 1.5 times the upper limit of normal value (ULN); AST and alt ≤ 5 times ULN; Serum total bilirubin (TBIL) ≤ 1.5 times ULN; International normalized ratio (INR) ≤ 1.5 times ULN, or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN (except for patients undergoing anticoagulant therapy);
11. Male patients and female subjects of childbearing age should agree to take effective contraceptive measures from the signing of informed consent to 3 months after the last administration;
12. Patients with herpes need 3 months after the end of herpes treatment.

Exclusion Criteria:

1. Patients with a history of primary uveal melanoma or any other (including unknown primary) malignancy within 5 years before the first administration of the trial treatment.

   Note: 1 or 2 stage skin basal / squamous cell carcinoma, superficial bladder cancer or orthotopic carcinoma receiving potentially curative treatment are the most effective treatments;
2. Liver lesions are not suitable for intratumoral injection or do not meet the injection volume requirements;
3. Patients who had received anti herpes simplex virus treatment within 4 weeks before the first administration of the trial treatment, such as acyclovir, ganciclovir, valacyclovir, arabine adenosine, etc;
4. Patients with active or history of autoimmune diseases that may recur (such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulitis, etc.), or patients with high risk (such as organ transplantation and immunosuppressive treatment). However, subjects with the following diseases are allowed to be included in the group:

   * stable type 1 diabetic patients after a fixed dose of insulin.
   * autoimmune hypothyroidism or Hashimoto's thyroid inflammation requiring only hormone replacement therapy;
   * skin diseases that do not require systemic treatment (such as eczema, skin rash accounting for less than 10% of the body surface, psoriasis without ophthalmic symptoms, etc.);
   * celiac disease that has been controlled;
   * any other disease that will not recur without external inducing factors;
5. Patients with major surgery are expected to include a 28 day screening period during the study period;
6. Patients requiring systemic corticosteroids (equivalent to > 10mg prednisone / day) or other immunosuppressive drugs within 14 days before enrollment or during the study. However, you are allowed to join the group under the following conditions:

   * subjects were allowed to use topical or inhaled glucocorticoids;
   * allow short-term (≤ 7 days) use of glucocorticoids to prevent or treat non autoimmune allergic diseases;
7. Patients with active gastrointestinal ulcer, incomplete intestinal obstruction, active gastrointestinal bleeding and perforation;
8. Patients suffering from interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung disease, acute radiation pneumonia, etc;
9. Uncontrolled stable systemic diseases such as cardiovascular and cerebrovascular diseases, hypertension, diabetes, tuberculosis and so on.
10. History of infection with human immunodeficiency virus, or suffer from other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation or stem cell transplantation;
11. patients with hepatitis B surface antigen (HBsAg) positive and hepatitis B virus (HBV) DNA copy number >1x103 copy /mL;
12. Patients with hepatitis C virus (HCV) antibody positive or human immunodeficiency virus (HIV) antibody positive;
13. Patients with severe infection within 4 weeks before the first administration, or patients with active infection requiring intravenous antibiotic treatment within 2 weeks before the first administration, and patients with unexplained fever > 38.5 ℃ before the first administration;
14. Patients known to have severe allergic reactions to herpes virus, macromolecular protein preparation / monoclonal antibody, or any known test drug components (CTCAE v5.0 grade is greater than grade 3);
15. Participated in clinical trials of other drugs within 4 weeks before the first administration;
16. Alcohol addicts or have a history of drug abuse or drug abuse in recent 1 year;
17. Having a clear history of neurological or mental disorders, such as epilepsy, dementia, poor compliance, or peripheral nervous system disorders;
18. Pregnant or lactating women;
19. Patients who received live attenuated vaccine within 30 days before the first administration;
20. The researchers believe that patients who are not suitable to participate in the trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR(6 months) | From first dose up to 6 months, approximately.
  ORR(6 month) is defined as the proportion of subjects with complete response (CR) and partial response (PR) after 6 months of treatment.

SECONDARY OUTCOMES:
DCR(6 months) | Time Frame: From first dose up to 6 months, approximately.
  DCR(6 month) is defined as the proportion of subjects with complete response (CR) , partial response (PR) and stable disease(SD) after 6 months of treatment.
PFS | From first dose up to 12 months, approximately.
  PFS is defined as the time from the beginning of treatment to tumor progression or death from any cause.
OS | From first dose up to 12 months, approximately.
  OS is defined as the time from the beginning of treatment to death due to any cause.
overall survival rate（one year） | From first dose up to 12 months, approximately.
  defined as the proportion of patients who survived after 1 year of treatment
overall survival rate（two years） | From first dose up to 24 months, approximately.
  defined as the proportion of patients who survived after 2 year of treatment

IPD SHARING:
Plan to Share IPD: No